CLINICAL TRIAL: NCT01261507
Title: Reader Study to Demonstrate That Use of DeltaView™ is Superior to the Use Standard Prior and Current Antero/Posterior (AP/PA) X-ray Image Pair
Brief Title: Reader Study of DeltaView™ Chest Radiograph Software
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: Riverain Medical Group, Miamisburg, OH (Unknown); BioStat Solutions, Inc., Mt. Airy, MD (Industry)
Responsible Party: Principal Investigator, Matthew T. Freedman, MD, Associate Professor Oncology, Georgetown University
Other Study IDs: DHF-183-0531A
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Lung Neoplasm
Keywords: lung neoplasm nodule image processing computer-assisted
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
A new software product takes two chest radiographs, aligns them, and then subtracts one image from the other. The resulting image represents an image showing any differences between them. The study is to determine whether radiologists using this new software perform better with it than when they do not use it.

ELIGIBILITY:
Inclusion Criteria:

For Radiologists: American Board of Radiology Certification and live within the Baltimore, MD-Washington, DC Metropolitan areas

For chest radiographs, evidence of the presence or absence of lung nodule confirmed by expert panel; adequate image quality

-

Exclusion Criteria:

Radiologists who assisted by providing cases for review

For chest radiographs: poor image quality

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Radiologists in community practice of radiology chest radiographs of individuals with or without a lung nodule
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T Freedman, MD, MBA, Principal Investigator — Georgetown University; S.-C. Ben Lo, PhD, Principal Investigator — Georgetown University
Locations (1):
- ISIS Research Center, Georgetown University Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited by email 15 radiologists practicing in the DC Metro area. Used prior subjects and those referred by prior research subjects.
Pre-assignment Details: discussion of project was done with each participant. Any questions were answered and signed consent was obtained. There were no dropouts of those recruited.
Groups:
- Board Certified Radiologists: 15 Board Certified radiologists were recruited from non-University sites. Each served as subject and control is a crossover design
Period: Overall Study
Arm/Group | Board Certified Radiologists
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Radiologists: Board Certified Radiologists working in the Washington, DC, Baltimore region
Arm/Group | Radiologists
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants] — Radiologists interpretations without use of tested software
  Participants
    <=18 years | 0
    Between 18 and 65 years | 15
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Localized Receiver Operating Characteristic (LROC) Comparison
Description: The area under the LROC curve will be compared for the chest radiograph interpretations done without the new software and those done with the new software. Improvement will be demonstrated if the improvement with the new software is statistically significant at the p=<0.05. There were 422 cases in the total study. 20 of these were inserted as "noise" cases, not to be analyzed. Thus there were 402 cases to be analyzed. There were 120 cases with nodules and 282 without a nodule. LROC is a method for measuring the success or failure of a method where there is a tradeoff between the detection of lung nodules that are there (true positives) and the detection that the radiologist considers to be a nodule where no nodule is present (false positive). It yields a single number that done not have a unit of measurement.
Time Frame: 1 day
Population: All participants were included for calculation of A-LROC and Sensitivity-Specificity. All radiographs were interpreted both without and with software assistance
Measure: Mean (Standard Error); unit: unitless
Units Other Than Participants: responses on radiographs
Groups:
- Board Certified Radiologists Working Without Software: 15 Board Certified radiologists were recruited from non-University sites. Each served as subject and control is a crossover design
- Radiologists Working With Software: Each radiologist serves as own control, working without and with software. This is the arm working with software
Arm/Group | Board Certified Radiologists Working Without Software | Radiologists Working With Software
Number analyzed (Participants) | 15 | 15
Number analyzed (responses on radiographs) | 402 | 402
unitless | 0.477 (0.037) | 0.536 (0.037)
Statistical Analysis 1: Comparison: Board Certified Radiologists Working Without Software vs Radiologists Working With Software; Measure is the difference between the radiologists working without the software less the value for the radiologists working with the software. Thus a negative value would indicate that the the radiologists showed better results when using the software; Test type: Superiority or Other; p < 0.05, mixed model:Dorfman, Berbaum, Metz; difference in areas under the LROC curve = -0.059, 95% CI 2-sided [-0.086 to -0.031], Standard Error of Mean 0.037

2. Secondary Outcome: Sensitivity and Specificity
Description: Sensitivity and specificity will be measured. If the radiologists using the new software have higher sensitivity, statistically significant at the p=< 0.05, the use of the new software will be considered to have resulted in improvement. A decrease in specificity is expected.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: Percentage of cases
Groups:
- Radiologists Working Without Software: Radiologists interpret the same images without the use of software
- Radiologists Working With Software: radiologists interpret the images using the experimental software
Arm/Group | Radiologists Working Without Software | Radiologists Working With Software
Number analyzed (Participants) | 15 | 15
Percentage of cases
  Sensitivity: correct detection of cancer | 43.8 (0.36) [0.092 to -0.033] | 50.1 (0.36) [0.092 to -0.033]
  Specificity: cancer free cases correctly identifie | 94.1 (0.12) | 92.6 (0.12)

3. Secondary Outcome: False Positive Decisions of Radiologists
Description: This is a comparison of the radiologists working without and with the software. The false positive rate is the percentage of cases in which the radiologists identified a lesions/location suspected of being cancer at a location where cancer was not present. . A false positive represents a location selected on a chest image without cancer and, also, a mark on a chest image where cancer was present, but a different location, one without cancer, was marked.The radiologists could mark up to five locations on an image and had to provide a confidence rating for each. This analysis is of the single mark with the highest confidence level.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: percentage of marks not on cancers
Arm/Group | Radiologists Working Without Software | Radiologists Working With Software
Number analyzed (Participants) | 15 | 15
percentage of marks not on cancers | 9.7 (1.9) | 11.2 (1.9)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Board Certified Radiologists
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
The main limitation is that the experimental format for this study is similar to, but not identical to the clinical pattern of practice in that more data is recorded during the study than would normally be gathered in clinical practice

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less